CLINICAL TRIAL: NCT03289585
Title: Development and Maintenance of a National Registry For Patients With Hidradenitis Suppurativa
Brief Title: A National Registry For Patients With Hidradenitis Suppurativa
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-3835 (AECOM)
Record Dates: First submitted 2017-09-11; First posted 2017-09-21 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa; Registry
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hidradenitis Suppurativa Cohort: Patients with Hidradenitis Suppurativa (ages 18-99 years old) will be asked to complete a series of questionnaires on how Hidradenitis Suppurativa impacts quality of life.

SUMMARY:
The goal of this study is to get a better understanding of the skin condition, Hidradenitis Suppurativa, and to find out how the disease affects quality of life. The investigators hope this information will help improve treatment for this skin condition.

DETAILED DESCRIPTION:
The goal of this study is to get a better understanding of the skin condition, Hidradenitis Suppurativa, and to find out how the disease affects quality of life. The investigators will utilize a compilation of validated questionnaires including the Beck Depression Inventory form, Dermatology Life Quality Index (DLQI), Skindex, SF-36 health survey, the Quality of Life Enjoyment and Satisfaction Questionnaire- short form (Q-LES-Q-SF) and the Employment/Productivity Health Economic Questionnaire as well as other relevant clinical data. The investigators will additionally collect a modified Hidradenitis Suppurativa Lesion, Area, and Severity Index (HS-LASI) (or other appropriate disease severity score as determined by the team) from the physician of each enrollee. The investigators hope this information will help improve treatment for this skin condition.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18-99 years of age who have a diagnosis of Hidradenitis Suppurativa (as deemed by a physician at the Montefiore Hidradenitis Suppurativa Treatment Center)

Exclusion Criteria:

* Patients without a diagnosis of Hidradenitis Suppurativa or under the age of 18
* Patients who are unable to answer given questions within the 6 surveys
* Patient who are unable to be clinically evaluated by a Montefiore physician

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy adults (ages 18-99) with a diagnosis of Hidradenitis Suppurativa
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
Skin-related quality of life | Baseline
  Quality of life as measured using standardized Dermatology Quality of Life Index
Presence and severity of depression | Baseline
  Presence and severity of depression as measured using standardized Beck Depression Inventory
Skin-related of life | Baseline
  Quality of life as measured using standardized SkinDex questionnaires
Subject-reported subject health | Baseline
  Subject-reported subject health as measured using the standardized SF-36 questionnaires
Degree of enjoyment and satisfaction experienced by subjects in daily functioning. | Baseline
  Degree of enjoyment and satisfaction experienced by subjects in various areas of daily functioning as measured by the standardized Quality of Life Enjoyment and Satisfaction Questionnaire-short form.
Employment and economic productivity | Baseline
  Self-reported employment and economic productivity as measured by a standardized health economic questionnaire

SECONDARY OUTCOMES:
Change in quality of life | At 6 months
  Change in quality of life as measured using standardized Dermatology Quality of Life Index after treatment initiation
Change in presence and severity of depression | At 6 months
  Change in presence and severity of depression as measured using standardized Beck Depression Inventory after treatment initiation
Change in quality of life | At 6 months
  Change in quality of life as measured using standardized SkinDex questionnaires after treatment initiation
Change in subject-reported subject health | At 6 months
  Change in subject-reported subject health as measured using standardized SF-36 questionnaires after treatment initiation
Change in degree of enjoyment and satisfaction experienced by subjects in various areas of daily functioning | At 6 months
  Change in degree of enjoyment and satisfaction experienced by subjects in various areas of daily functioning as measured by the standardized Quality of Life Enjoyment and Satisfaction Questionnaire-short form after treatment initiation
Change in self-reported employment and economic productivity | At 6 months
  Change in self-reported employment and economic productivity as measured by a standardized health economic questionnaire after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Cohen, MD, MPH, Principal Investigator — Albert Einstein College of Medicine Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data to other researchers

REFERENCES:
- See also: Montefiore Hidradenitis Suppurativa Multispecialty Treatment Center — http://www.montefiore.org/hidradenitis-suppurativa